CLINICAL TRIAL: NCT01676467
Title: A Sample Collection Protocol for Disease Profiling of Smoking Asthma.
Brief Title: Sample Collection in Smoking Asthma
Status: Completed | Type: Observational
Sponsor: Respivert Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: ENA002
Record Dates: First submitted 2012-08-21; First posted 2012-08-31 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Smoking asthma on steroids: Smokers with persistent asthma on background steroid therapy
- Smoking asthma steroid naïve: Smokers with persistent asthma, steroid naive
- asthma on steroids: Non-Smokers with persistent asthma on background steroid therapy
- asthma, steroid naïve: Non-smokers with persistent asthma, steroid naive
- Healthy smoking: Healthy smoking control subjects
- Healthy non-smoking: Healthy non-smoking control subjects

SUMMARY:
This study will collect blood and sputum (phlegm) samples from subjects with asthma, smokers and normal healthy subjects, to compare the biological markers of disease and inflammation.

ELIGIBILITY:
Inclusion Criteria (healthy subjects):

* Male or female, between 18 and 55 years of age, inclusive.
* no clinically significant abnormalities.
* able to produce an adequate induced sputum sample.
* no history of chronic respiratory disease including asthma.
* no history of allergic symptoms e.g., allergic rhinitis, eczema.
* No other acute illness in the 6 weeks prior to Visit 1.

Additional Inclusion Criterion for Healthy Smoking Subjects

* Be a smoker for >/= 1 year.

Additional Inclusion Criteria (Persistent Asthmatic Subjects):

* No contraindications to the procedures in this study.
* Symptoms compatible with asthma for at least 6 months prior to screening
* Pre-bronchodilator FEV1 >/=50% predicted at Visit 1.
* clinically stable asthma for at least 6 weeks prior to Visit 1.
* No acute illness including asthma exacerbation requiring augmentation of therapy in the 6 weeks prior to Visit 1.
* on current asthma controller therapy for >/= 6 weeks prior to Visit 1.

Additional Inclusion for Steroid Naïve Asthmatics (smoking or non-smoking)

* Must not have received a regular course of inhaled or oral corticosteroids for at least 3 months prior to Visit 1.

Additional Inclusion for Smoking Asthmatics

* Be a smoker for >/= 1 year prior to Visit 1.

Exclusion Criteria (healthy):

* History of any clinically significant medical illness or medical disorders.
* Diagnosis of chronic obstructive pulmonary disease (COPD), cystic fibrosis, or other significant respiratory disorder including significant occupational or environmental exposures with ongoing respiratory symptoms.
* bronchodilator response of >/=12% and at least 200 mL from baseline or an FEV1 value <85% of predicted value at Visit 1.
* positive urine pregnancy screening result.
* recent history (within previous 6 months) of alcohol or drug abuse.
* Positive urine toxicology screen for substances of abuse
* positive serology test for HIV antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (anti-HCV) at Visit 1.
* Received an experimental antibody or biologic therapy within the 6 months prior to Visit 1, or received any other experimental therapy or new investigational agent within 60 days of Visit 1.
* Is an employee or family member of the investigator, study centre or Sponsor.
* Any condition that, in the opinion of the investigator, would complicate or compromise the study, or the well-being of the subject.
* Use of any antioxidants within 1 week of Visit 1 and throughout the study period.
* known allergies, hypersensitivity, or intolerance to short acting β-agonists (SABA).

Additional Exclusion Criterion for Healthy Non-smoking Subjects

* subject is a smoker (regular or irregular), or has smoked or used nicotine-containing products within the 6 months prior to Visit 1.

Additional Exclusion Criteria (Persistent Asthma Subjects):

* Diagnosis of allergic bronchopulmonary aspergillosis (ABPA), allergic bronchopulmonary mycosis (ABPM), or occupational asthma.
* Diagnosis of COPD, cystic fibrosis, or other significant respiratory disorder including significant occupational or environmental exposures with ongoing respiratory symptoms.
* Use of theophylline, N-acetyl cysteine, or any other anti-oxidants within 1 week of Visit 1 and throughout the study period.
* positive test for tuberculosis at Visit 1.

Additional Exclusion Criterion for Non-smoking Asthmatic Subjects

* subject is a smoker (regular or irregular), or has smoked or used nicotine-containing products within the 6 months prior to Visit 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be selected by advertisements from the general population and primary care.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Sputum and serum biomarkers | Day 10
  Measurement of biomarkers of inflammation, including but not limited to: TNFα, IL-8, IFNγ, IP10 and eotaxin in sputum supernatant and serum will be collected and measured only once, at Visit 2 (Day 10).
Sputum cell count | Day 10
  Sputum cell count (total cells, differentials and absolute number) at Visit 2 (Day 10).

CONTACTS AND LOCATIONS:
Overall Officials: Dr Garth Rapeport, Study Director — Respivert Ltd
Locations (1):
- Harrow, Middlesex, United Kingdom